CLINICAL TRIAL: NCT07182110
Title: Effect of Dexamethasone-Enhanced TAP Block Mixture on Postoperative Analgesia in Laparoscopic Cholecystectomy
Brief Title: Dexamethasone-Enhanced TAP Block in Lapchole
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Mohamad-Ali Barada, Anesthesia Attending, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MGH-07-25037
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Transversus Abdominis; Nerve Block; Dexamethasone; Pain; Acute Pain; Pain Management; Breakthrough Pain; Analgesics, Opioid; Anesthesia
MeSH Terms: conditions — Pain; Acute Pain; Agnosia; Breakthrough Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Marcaine (Active Comparator)
  Interventions: Drug: Marcaine- 0.25%
- Marcaine and Dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone enhanced TAP Block

INTERVENTIONS:
Drug: Dexamethasone enhanced TAP Block — 20 ml Marcaine containing 0.25% bupivacaine + 4 mg dexamethasone + normal saline
  Arms: Marcaine and Dexamethasone
Drug: Marcaine- 0.25% — 20 ml solution containing 0.25% bupivacaine + normal saline
  Arms: Marcaine

SUMMARY:
The transversus abdominis plane (TAP) block is widely used as part of analgesia for abdominal surgeries such as laparoscopic cholecystectomy. While bupivacaine is commonly used for TAP blocks with reported success. Dexamethasone is often used as an adjuvant in prolonging duration of blocks; however, data on its efficacy in enhancing TAP blocks in laparoscopic cholecystectomy remain limited. This study aims to assess whether adding dexamethasone to bupivacaine in a TAP block improves postoperative pain control and reduces opioid consumption

DETAILED DESCRIPTION:
Hypothesis Patients receiving a dexamethasone-enhanced TAP block will have a longer duration of analgesia, lower postoperative pain scores, and reduced opioid requirements compared to patients receiving local anesthetic alone.

Objectives

* Primary Objective:
* To evaluate the time to first postoperative analgesic request.
* Secondary Objectives:
* To assess postoperative pain using the Visual Analog Scale (VAS).
* To evaluate the incidence of postoperative nausea and vomiting (PONV).
* To compare total postoperative analgesic consumption.
* To assess the need for rescue analgesia.

Methods Study Design

* Prospective, randomized, double-blind clinical trial. Study Population
* Adult patients (age ≥18), ASA physical status I to III, planned for elective laparoscopic cholecystectomy. Interventions
* All patients will undergo standard general anesthesia.
* TAP block will be performed pre-induction bilaterally by an experienced anesthesiologist blinded to the injectate.
* Patients will be randomized into two groups:
* Group A (Control): 20 ml solution containing 0.25% bupivacaine + normal saline
* Group B (Intervention): 20 ml solution containing 0.25% bupivacaine + 4 mg dexamethasone + normal saline

All patients will receive standard postoperative care, including paracetamol and antiemetics

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients
* Laparoscopic Cholecystectomy Patients
* Patients able to consent

Exclusion Criteria:

* Patients allergic to dexamethasone
* Allergic to Marcaine
* Hemodynamically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Time to first analgesic requirement (in hours) | within 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Makassed General Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghani SA, Hussain HU, Wahid MA, Majeed N, Burney S, Tanveer A, Asghar MS. Laparoscopic-assisted versus ultrasound-guided transversus abdominis plane block for laparoscopic cholecystectomy: a systematic review and meta-analysis. BMC Surg. 2024 Dec 21;24(1):400. doi: 10.1186/s12893-024-02706-7. PMID 39709396
- [Background] Uzunay NT, Mingir T, Erginoz E, Karakas DO, Kose E. Comparison of laparoscopic-guided versus ultrasound-guided TAP block in laparoscopic cholecystectomy. Cir Cir. 2024;92(2):174-180. doi: 10.24875/CIRU.23000394. PMID 38782390
- [Background] Taheri P, Moinfar Z, Varpaei HA. Comparison of the Stress Responses After TAP Block and Epidural Anesthesia in Patients Undergoing Elective Laparoscopic Cholecystectomy Under General Anesthesia: Randomized Clinical Trial. Clin J Pain. 2023 Jul 1;39(7):319-325. doi: 10.1097/AJP.0000000000001117. PMID 37083674
- [Background] Nair P, Behera CR, Patra RK, Shekar N, Rao LS, Pujari P, Panda B, Mishra A. Efficacy and Cost-Effectiveness of Laparoscopic Transversus Abdominis Plane (TAP) Block in Laparoscopic Cholecystectomy: A Comparison With the Non-TAP Group. Cureus. 2022 Nov 30;14(11):e32038. doi: 10.7759/cureus.32038. eCollection 2022 Nov. PMID 36600856